CLINICAL TRIAL: NCT00000818
Title: Evaluation of the Changes in HIV-1 Burden in Peripheral Blood and Lymphoid Tissue Following Zidovudine ( AZT ) Treatment in HIV-1-Infected Patients With CD4+ Cells Between 100 and 500 Cells/mm3.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: DATRI 012
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-07-29 (Estimated); Status verified 1996-05

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine; Lymph Nodes; Lymphoid Tissue
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
PRIMARY: To determine the effect of 8 weeks of zidovudine (AZT) treatment on the HIV-1 burden in peripheral blood and lymphoid tissue in HIV-1-infected, AZT-naive patients with CD4+ T lymphocyte counts between 100 and 500 cells/mm3.

SECONDARY: To determine the extent to which apoptosis (programmed cell death) occurs in these patients.

In previous trials of AZT treatment in HIV-infected patients, an antiviral effect has been clearly demonstrated by quantitative measurement of virus in plasma and peripheral blood mononuclear cells. However, the lymphoid tissues appear to be a major reservoir for HIV-1 and a major site of virus replication in HIV-infected persons. Further data is needed to assess the effect of treatment on viral burden and HIV-1 replication in lymphoid tissue.

DETAILED DESCRIPTION:
In previous trials of AZT treatment in HIV-infected patients, an antiviral effect has been clearly demonstrated by quantitative measurement of virus in plasma and peripheral blood mononuclear cells. However, the lymphoid tissues appear to be a major reservoir for HIV-1 and a major site of virus replication in HIV-infected persons. Further data is needed to assess the effect of treatment on viral burden and HIV-1 replication in lymphoid tissue.

Patients receive AZT daily for 8 weeks and are followed in clinic at weeks 2, 4, 6, 8, 9, and 14 (or possibly via telephone call at week 14). Patients undergo a lymph node biopsy at day 0 and week 8.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Prophylaxis against AIDS-related opportunistic infections.
* Supportive therapies, such as medications for nausea, vomiting, anemia, and analgesia.

Patients must have:

* HIV infection.
* CD4 count 100 - 500 cells/mm3.
* At least two palpable lymph nodes.
* Plasma viremia.
* No CURRENT AIDS-defining conditions.
* No prior antiretroviral treatment.

Exclusion Criteria

Concurrent Medication:

Excluded during the first 8 weeks of study:

* Other antiretroviral agents.
* Steroids.
* Interleukins.
* Interferons.
* Cytotoxic chemotherapy.

Prior Medication:

Excluded:

* Prior antiretroviral therapy.
* Prior cytotoxic chemotherapy.
* Acute therapy for an infection or another medical illness within 14 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18

CONTACTS AND LOCATIONS:
Overall Officials: Cohn J, Study Chair; Bilello J, Study Chair
Locations (9):
- United States (9):
  - Cedars Sinai Med Ctr, Los Angeles, California
  - Palo Alto Veterans Affairs Health Care System, Palo Alto, California
  - AIDS Community Research Consortium, Redwood City, California
  - Mount Zion Med Ctr / UCSF, San Francisco, California
  - North Broward Hosp District, Fort Lauderdale, Florida
  - Goodgame Med Group, Maitland, Florida
  - Univ of Illinois, Chicago, Illinois
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - Baylor College of Medicine / Houston Veterans Adm Med Ctr, Houston, Texas